CLINICAL TRIAL: NCT02982616
Title: Influence of Intragastric Fatty Acid Infusion on Behavioral Responses to Positive Emotion Induction in Normal Weight Subjects
Brief Title: Influence of Intragastric Fatty Acid Infusion on Behavioral Responses to Positive Emotion Induction in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S55863
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — lauric acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- positive emotion and fatty acid (Experimental): positive emotion induction combine with 2.g Dodecanoic acid intragastric infusion
  Interventions: Dietary Supplement: Dodecanoic acid; Behavioral: Positive emotion
- neutral emotion and fatty acid (Experimental): neutral emotion induction combine with 2.g Dodecanoic acid intragastric infusion
  Interventions: Dietary Supplement: Dodecanoic acid; Behavioral: neutral emotion
- positive emotion and saline (Experimental): positive emotion induction combine with saline intragastric infusion
  Interventions: Behavioral: Positive emotion; Dietary Supplement: saline
- neutral emotion and saline (Placebo Comparator): neutral emotion induction combine with saline intragastric infusion
  Interventions: Dietary Supplement: saline; Behavioral: neutral emotion

INTERVENTIONS:
Dietary Supplement: Dodecanoic acid — The middle chain saturated fatty acid that can be widely found in daily food.
  Other Names: Lauric acid
  Arms: neutral emotion and fatty acid; positive emotion and fatty acid
Behavioral: Positive emotion — Positive emotion induced by facial expressions and classic music.
  Arms: positive emotion and fatty acid; positive emotion and saline
Dietary Supplement: saline — saline
  Arms: neutral emotion and saline; positive emotion and saline
Behavioral: neutral emotion — Neutral emotion induced by facial expressions and classic music.
  Arms: neutral emotion and fatty acid; neutral emotion and saline

SUMMARY:
The purpose of this study is to test whether intragastrically infused fatty acid will interact with positive emotion induction and if this effect is mediated by gut hormones.

DETAILED DESCRIPTION:
This study aims at the possible effect of subliminal intragastric administration of fatty acids on responses to positive emotion induction, based on our earlier findings that subjective administration of fatty acid decreases neural responses to negative mood induction (Van Oudenhove et al, J Clin Invest 2011). After screening for exclusion criteria and the participants sign the informed consent form, an intravenous catheter is placed in the forearm, and a naso-gastric tube inserted through the nose. Then the test subject is connected to the equipment in order to record the activity of the autonomic nervous system, via three electrocardiogram electrodes. By using the nasogastric tube we serve a fatty acid solution (Dodecanoic acid, "fatty acid" condition) or a physiological saline solution ( "control" condition) intragastrically. The intragastric administration of low doses of this food ingredient has already been used in several previous studies by our research group and has proven perfectly safe. A positive or neutral emotional state will be induced by the combination of looking at emotional facial expressions and listening to classical music pieces that were previously validated for this purpose; This combination of incentives has already been used in previous studies of our research group. Responses will be measured by means of validated self-report scales and measurements of the vagal tone. We also take blood samples on a regular basis by the intravenous catheter for determination of gastrointestinal hormones, given our hypothesis that this may explain the effect on emotions. After removal of the nasogastric tube, the influence of subliminal administration of fatty acids and emotional state on food intake measured by means of a validated and previously drink test used in which participants "ad libitum" to drink a chocolate milkshake while the emotion-induction by means of classical music pieces continue. Finally, the intravenous catheter is removed.

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* age > 18 and < 60.
* Body Mass Index (BMI) of 19-25 kg/m2 (no weight change of more than 5% of body weight in the past three months).

Exclusion Criteria:

* chronic medical illness affecting the gastrointestinal, endocrine, cardiovascular or nervous system (risk of) pregnancy history of upper gastrointestinal surgery history of behavioral, therapeutic or surgical treatment aiming at or leading to weight loss/gain psychiatric disorders, including (history of) depression or eating disorders alcohol abuse or dependence regular use of medication, except for oral contraception use of any drugs, including cannabis, during the past 6 months

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
time evolution of VAS from the beginning until the end of a study visit | -10min 0min 10min 20min 30min 40min
  visual analogue scale for appetite related sensations
time evolution of gut hormones from the beginning until the end of a study visit | -10min 10min 20min 30min 40min

SECONDARY OUTCOMES:
evolution of heart rate variability | -20min 20min
hedonic food intake | 40min
  amount of milkshake drunk

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, Prof, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
Due to ethical rules the individual participant data will be kept confidential.

REFERENCES:
- [Background] Van Oudenhove L, McKie S, Lassman D, Uddin B, Paine P, Coen S, Gregory L, Tack J, Aziz Q. Fatty acid-induced gut-brain signaling attenuates neural and behavioral effects of sad emotion in humans. J Clin Invest. 2011 Aug;121(8):3094-9. doi: 10.1172/JCI46380. Epub 2011 Jul 25. PMID 21785220
- [Background] Parker BA, Sturm K, MacIntosh CG, Feinle C, Horowitz M, Chapman IM. Relation between food intake and visual analogue scale ratings of appetite and other sensations in healthy older and young subjects. Eur J Clin Nutr. 2004 Feb;58(2):212-8. doi: 10.1038/sj.ejcn.1601768. PMID 14749739
- [Background] Mayer EA. Gut feelings: the emerging biology of gut-brain communication. Nat Rev Neurosci. 2011 Jul 13;12(8):453-66. doi: 10.1038/nrn3071. PMID 21750565
- [Background] Mayer EA, Naliboff BD, Craig AD. Neuroimaging of the brain-gut axis: from basic understanding to treatment of functional GI disorders. Gastroenterology. 2006 Dec;131(6):1925-42. doi: 10.1053/j.gastro.2006.10.026. No abstract available. PMID 17188960
- [Background] Mitterschiffthaler MT, Fu CH, Dalton JA, Andrew CM, Williams SC. A functional MRI study of happy and sad affective states induced by classical music. Hum Brain Mapp. 2007 Nov;28(11):1150-62. doi: 10.1002/hbm.20337. PMID 17290372
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Derived] Zhao D, Boey L, Weltens N, Biesiekierski JR, Iven J, Depoortere I, Tack J, Van Oudenhove L. Influence of subliminal intragastric fatty acid infusion on subjective and physiological responses to positive emotion induction in healthy women: A randomized trial. Psychoneuroendocrinology. 2019 Oct;108:43-52. doi: 10.1016/j.psyneuen.2019.06.010. Epub 2019 Jun 13. PMID 31226660